CLINICAL TRIAL: NCT04382534
Title: A Cross-sectional and Cohort Study of COVID-19 Patients With Post - Discharge Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M20200421
Record Dates: First submitted 2020-04-26; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-04

CONDITIONS: Covid19; Respiratory Rehabilitation; Cross-sectional Study; Cohort Study
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rehabilitation guidance group: 1 to 2 times of rehabilitation instruction according to the rehabilitation instruction program, either online or in person.According to the rehabilitation instruction, the patient performed self-rehabilitation exercises in the isolation point.
- Systematic rehabilitation treatment: According to the systematic rehabilitation treatment program, the rehabilitation therapist entered the home for one-to-one rehabilitation treatment, once a day, for a total of 10 days.
  Interventions: Combination Product: Respiratory rehabilitation

INTERVENTIONS:
Combination Product: Respiratory rehabilitation — Health education and energy saving techniques, chest activity training, local lung dilation techniques, breathing training, airway clearance training, aerobic exercise, resistance training
  Groups: Systematic rehabilitation treatment

SUMMARY:
Post-discharge rehabilitation regimens for covid-19 patients have not been supported by high-quality evidence-based medical evidence.The first part of this study is a cross-sectional study.The contents of the study were the factors related to the dysfunction of COVID - 19 patients after discharge from the hospital in Wuhan.The second part of this study is a cohort study.To observe the functional changes of COVID-19 patients after discharge in hospital rehabilitation, home rehabilitation and no rehabilitation, in order to propose a more safe and effective rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* patients with definite diagnosis of COVID-19 normal or severe
* patients who entered the isolation point <3 days after discharge
* 18-80 years old
* agree to join the queue

Exclusion Criteria:

* body temperature >38°C
* heart rate >120 times/min or <40 times/min, systolic blood pressure <90mmHg or >180mmHg, respiratory rate >25 times/min in calm state.Or above vital signs fluctuate significantly.
* continuous oxygen therapy is required.
* patients with myocarditis, pulmonary hypertension, congestive heart failure, fresh venous thromboembolic diseases, unstable fractures and other inappropriate exercise
* patients with consciousness disorders, severe sequelae of cerebral infarction, cognitive dysfunction, mental disorders, severe balance disorders, and severe bone and joint diseases, which affect evaluation and treatment
* other conditions that cannot be cooperated with rehabilitation treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COVID-19 after discharge
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms and signs | Ten days
  To take a history and physical examination
Respiratory function | Ten days
  To take a physical examination and mMRC
The body function | Ten days
  To take a MMT, 6-min walking test and Borg Index
ADL | Ten days
  To take a modified Barthel index

CONTACTS AND LOCATIONS:
Locations (1):
- Huarunwugang general hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided